CLINICAL TRIAL: NCT00456365
Title: Effect of Statin Therapy on Disease Progression in Autosomal Dominant Polycystic Kidney Disease
Brief Title: Effect of Statin Therapy on Disease Progression in Autosomal Dominant Polycystic Kidney Disease (ADPKD)
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: University of Colorado, Denver (Other)
Collaborators: National Institute of Diabetes and Digestive and Kidney Diseases (NIDDK) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 05-0704; 2R01DK058793 (NIH)
Record Dates: First submitted 2007-03-12; First posted 2007-04-04 (Estimated); Results first posted 2018-03-09 (Actual); Last update posted 2018-03-09 (Actual); Status verified 2018-02

CONDITIONS: Polycystic Kidney, Autosomal Dominant
Keywords: Autosomal dominant polycystic kidney disease; Cystic kidney disease; High blood pressure; Statin
MeSH Terms: conditions — Polycystic Kidney, Autosomal Dominant; Kidney Diseases, Cystic; Hypertension | interventions — Pravastatin

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Pravastatin (Experimental): Pravastatin
  Interventions: Drug: pravastatin
- Placebo (Placebo Comparator): Placebo
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: pravastatin — Pravastatin 20 mg daily (subject age 8-12 years) or 40 mg daily (subject age 13-21 years)
  Arms: Pravastatin
Drug: Placebo — Placebo daily
  Arms: Placebo

SUMMARY:
The purpose of this study is to determine whether the medication pravastatin will ameliorate renal and cardiovascular disease over a 3-year period in children and young adults with autosomal dominant polycystic kidney disease (ADPKD).

DETAILED DESCRIPTION:
Autosomal dominant polycystic kidney disease (ADPKD) is the most common hereditary kidney disease, affecting 1 in 400 to 1000 individuals and accounting for 4% of end-stage renal disease in the United States and 8-10% in Europe. The condition is characterized by progressive development of kidney cysts with kidney enlargement and associated loss of kidney function. High blood pressure and cardiovascular disease are common in patients with ADPKD. Although the condition is often thought to affect primarily adults, it is clear that the disease can be present in the fetus and young children.

This study was designed to determine if treatment with the medicine pravastatin can slow the progression of kidney and heart disease when initiated early in life in patients with ADPKD. The Investigators will assess differences between pravastatin and placebo study groups over the three-year study period with respect to: 1) total kidney volume as assessed by magnetic resonance imaging (MRI); 2) left ventricular mass index as assessed by MRI; 3) urinary albumin excretion; and 4) endothelial-dependent vasodilation as assessed by brachial ultrasound. A total of 110 subjects were enrolled in this research study. This study involved pediatric subjects because the Investigators believe that early intervention is critical if they are to decrease the morbidity and mortality associated with this condition. If pravastatin is shown to be effective in ameliorating progression of renal and cardiovascular disease in this study, routine management of people with this condition will be drastically altered.

ELIGIBILITY:
Inclusion Criteria:

* Age 8-22 years
* Autosomal dominant polycystic kidney disease
* Normal kidney function

Exclusion Criteria:

* Abnormal kidney function
* Past allergic history to medications used in study
* Liver disease
* Muscle disease/dystrophy
* Pregnancy, planned pregnancy, or lactation within study period
* Inability to cooperate with or clinical contraindication for magnetic resonance imaging

Ages: 8 Years to 22 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 110 (Actual)
Dates: Start 2006-11; Primary Completion 2012-10 (Actual); Study Completion 2012-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Melissa A Cadnapaphornchai, MD, Principal Investigator — University of Colorado, Denver; Robert W Schrier, MD, Principal Investigator — University of Colorado, Denver
Locations (1):
- University of Colorado at Denver and Health Sciences Center, Denver, Colorado, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Schrier RW. Optimal care of autosomal dominant polycystic kidney disease patients. Nephrology (Carlton). 2006 Apr;11(2):124-30. doi: 10.1111/j.1440-1797.2006.00535.x. PMID 16669974
- [Background] Shamshirsaz AA, Reza Bekheirnia M, Kamgar M, Johnson AM, McFann K, Cadnapaphornchai M, Nobakhthaghighi N, Schrier RW. Autosomal-dominant polycystic kidney disease in infancy and childhood: progression and outcome. Kidney Int. 2005 Nov;68(5):2218-24. doi: 10.1111/j.1523-1755.2005.00678.x. PMID 16221221
- [Background] Taylor M, Johnson AM, Tison M, Fain P, Schrier RW. Earlier diagnosis of autosomal dominant polycystic kidney disease: importance of family history and implications for cardiovascular and renal complications. Am J Kidney Dis. 2005 Sep;46(3):415-23. doi: 10.1053/j.ajkd.2005.05.029. PMID 16129202
- [Background] Cadnapaphornchai MA, Fick-Brosnahan GM, Duley I, Johnson AM, Strain JD, DeGroff CG, Schrier RW. Design and baseline characteristics of participants in the study of antihypertensive therapy in children and adolescents with autosomal dominant polycystic kidney disease (ADPKD). Contemp Clin Trials. 2005 Apr;26(2):211-22. doi: 10.1016/j.cct.2005.01.001. PMID 15837441
- [Background] Fick-Brosnahan GM, Belz MM, McFann KK, Johnson AM, Schrier RW. Relationship between renal volume growth and renal function in autosomal dominant polycystic kidney disease: a longitudinal study. Am J Kidney Dis. 2002 Jun;39(6):1127-34. doi: 10.1053/ajkd.2002.33379. PMID 12046022
- [Background] Kelleher CL, McFann KK, Johnson AM, Schrier RW. Characteristics of hypertension in young adults with autosomal dominant polycystic kidney disease compared with the general U.S. population. Am J Hypertens. 2004 Nov;17(11 Pt 1):1029-34. doi: 10.1016/j.amjhyper.2004.06.020. PMID 15533729
- [Derived] St Pierre K, Cashmore BA, Bolignano D, Zoccali C, Ruospo M, Craig JC, Strippoli GF, Mallett AJ, Green SC, Tunnicliffe DJ. Interventions for preventing the progression of autosomal dominant polycystic kidney disease. Cochrane Database Syst Rev. 2024 Oct 2;10(10):CD010294. doi: 10.1002/14651858.CD010294.pub3. PMID 39356039
- See also: PKD Foundation website — http://www.pkdcure.org

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Pravastatin | Placebo
Started | 56 | 54
Completed | 49 | 42
Not Completed | 7 | 12
Not completed — Lost to Follow-up | 1 | 3
Not completed — Withdrawal by Subject | 4 | 7
Not completed — Pregnancy | 1 | 1
Not completed — oncologic diagnosis | 1 | 1

BASELINE CHARACTERISTICS:
Population: A total of 111 participants were screened with 110 enrolled in this clinical trial, including 56 randomized to pravastatin and 54 randomized to placebo.
Groups:
- Total: Total of all reporting groups
Arm/Group | Pravastatin | Placebo | Total
Number analyzed (Participants) | 56 | 54 | 110
Age, Continuous [Mean (Standard Deviation); unit: years] | 16 (4) | 16 (4) | 16 (4)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 34 | 34 | 68
  Male | 22 | 20 | 42
Region of Enrollment [Number; unit: participants]
  United States | 56 | 54 | 110
Total kidney volume corrected for height [Mean (Standard Deviation); unit: ml/m] — Total kidney volume corrected for height (HtTKV, ml/m)
  ml/m | 336 (187) | 315 (175) | 326 (181)
Urinary albumin excretion [Mean (Standard Deviation); unit: mcg/min] — Urinary albumin excretion in mcg/min
  mcg/min | 27 (37) | 51 (123) | 39 (79)
Left ventricular mass index [Mean (Standard Deviation); unit: g/m^2] — Left ventricular mass index in g/m^2 by MRI
  g/m^2 | 55 (12) | 53 (10) | 54 (11)
Total cholesterol [Mean (Standard Deviation); unit: mg/dL] | 145 (30) | 151 (27) | 148 (29)
LDL cholesterol [Mean (Standard Deviation); unit: mg/dL] | 84 (23) | 90 (21) | 86 (22)

OUTCOME MEASURES:

1. Primary Outcome: Percent of Participants Demonstrating 20% or More Increase in Total Kidney Volume
Description: Percent of participants demonstrating 20% or more increase in total kidney volume corrected for height, left ventricular mass index, or urinary albumin excretion over the three year study period
Time Frame: 3 years
Population: Intention to treat
Measure: Number; unit: percentage of participants
Arm/Group | Pravastatin | Placebo
Number analyzed (Participants) | 49 | 42
percentage of participants | 69 | 88
Statistical Analysis 1: Comparison: Pravastatin vs Placebo; Test type: Superiority or Other; p = 0.03, Chi-squared

2. Secondary Outcome: Percentage Change in Total Kidney Volume Corrected for Height
Time Frame: 3 years
Population: ITT
Measure: Mean (Standard Deviation); unit: Percent change
Arm/Group | Pravastatin | Placebo
Number analyzed (Participants) | 49 | 42
Percent change | 23 (3) | 31 (3)
Statistical Analysis 1: Comparison: Pravastatin; Test type: Superiority or Other; p = 0.02, ANCOVA

3. Secondary Outcome: Left Ventricular Mass Index
Description: left ventricular mass index in g/m^2 by MRI
Time Frame: 3 years
Measure: Mean (Standard Deviation); unit: g/m^2
Arm/Group | Pravastatin | Placebo
Number analyzed (Participants) | 49 | 42
g/m^2 | 60 (15) | 58 (13)
Statistical Analysis 1: Comparison: Pravastatin vs Placebo; Test type: Superiority or Other; p = 0.69, ANOVA

4. Secondary Outcome: Urinary Albumin Excretion
Time Frame: 3 years
Measure: Mean (Standard Deviation); unit: mcg/min
Arm/Group | Pravastatin | Placebo
Number analyzed (Participants) | 49 | 42
mcg/min | 29 (39) | 49 (99)
Statistical Analysis 1: Comparison: Pravastatin vs Placebo; Test type: Superiority or Other; p = 0.21, ANCOVA

ADVERSE EVENTS:
Arm/Group | Pravastatin | Placebo
Serious Adverse Events (participants affected / at risk) | 0/56 | 0/54
Other Adverse Events (participants affected / at risk) | 0/56 | 0/54

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No